CLINICAL TRIAL: NCT07283354
Title: Comparison of Acceleromyography and Electromyography in Obese Patients Undergoing General Anesthesia With Rocuronium: A Prospective Observational Study
Brief Title: Comparison of Acceleromyography and Electromyography in Obese Patients Undergoing General Anesthesia
Acronym: OBAEG
Status: Not yet recruiting | Type: Observational
Sponsor: University of Padova (Other)
Collaborators: University Hospital, Padua, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: AOP3692_CET; 6296/EST/25 (Other: Territorial Ethics Committee - Central-East Veneto Area)
Record Dates: First submitted 2025-11-25; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: Bariatric Surgery; General Anesthesia; Neuromuscular Blockade; Neuromuscular Monitoring; Acceleromyography; Electromyography
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with obesity undergoing bariatric surgery: Adults with obesity scheduled for bariatric surgery under general anesthesia. Each participant will be monitored for neuromuscular function using both acceleromyography (AMG) and electromyography (EMG) during surgery and after administration of sugammadex.
  Interventions: Procedure: Neuromuscular monitoring with electromyography (EMG); Procedure: Neuromuscular monitoring with acceleromyography (AMG)

INTERVENTIONS:
Procedure: Neuromuscular monitoring with electromyography (EMG) — Neuromuscular function will be assessed using an electromyography device applied to the hand. The device measures the electrical activity of muscles in response to ulnar nerve stimulation to calculate the Train-of-Four (TOF) ratio.
Procedure: Neuromuscular monitoring with acceleromyography (AMG) — Neuromuscular function will be assessed using an acceleromyography device applied to the hand. The device measures the acceleration of thumb movement in response to ulnar nerve stimulation to calculate the Train-of-Four (TOF) ratio.

SUMMARY:
The goal of this prospective observational study is to compare two different methods of monitoring muscle relaxation during anesthesia - acceleromyography (AMG) and electromyography (EMG) - in people with obesity who are having bariatric surgery with general anesthesia and the muscle relaxant rocuronium.

The main question is: Which method is more accurate and precise in measuring the Train-of-Four (TOF) ratio during surgery? As part of this comparison, researchers will also note how quickly each method detects recovery of muscle function after the reversal drug sugammadex.

Participants will:

* Receive standard anesthesia care for bariatric surgery, including rocuronium to relax the muscles.
* Have two small monitoring devices applied, one to each hand: AMG on one hand, EMG on the other.
* Be monitored for muscle function during surgery and after receiving sugammadex to reverse the muscle relaxation.

Researchers will also record how easy each device is to use and whether participants have any breathing problems after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Pathological obesity (Class II with comorbidities or Class III)
* Scheduled for bariatric surgery under general anesthesia
* Written informed consent obtained

Exclusion Criteria:

* Severe acute or chronic respiratory disease (e.g., asthma, COPD, severe restrictive disease)
* Severe acute or recent cardiac disease (e.g., acute or recent myocardial infarction, inducible ischemia, heart failure)
* End-stage hepatic or renal disease
* Intolerance, allergy, or contraindication to study-related drugs
* Absence of informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-65 years with pathological obesity (Class II with comorbidities or Class III) scheduled for bariatric surgery under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean paired difference in TOF ratio (AMG vs EMG) | Intraoperative period
  Mean difference between acceleromyography (AMG) and electromyography (EMG) measurements of the Train-of-Four (TOF) ratio (unitless) obtained from paired intraoperative recordings.

SECONDARY OUTCOMES:
Time to optimal conditions for tracheal intubation | From rocuronium administration to tracheal intubation (approximately 1-3 minutes).
  Time from rocuronium administration to achievement of optimal intubation conditions, defined as TOF count = 0 or deep block confirmed by post-tetanic count (PTC). Measured with both AMG and EMG.
Maintenance of deep neuromuscular block | From induction of anesthesia to start of reversal with sugammadex (approximately 60-120 minutes)
  Duration and stability of deep block (PTC < 5) maintained during anesthesia, as measured by AMG and EMG.
Time to recovery of TOF ratio ≥ 0.9 after sugammadex | From administration of sugammadex to achievement of TOF ratio ≥ 0.9 (typically 1-5 minutes).
  Time from administration of sugammadex to achievement of TOF ratio ≥ 0.9 with each monitoring method (AMG and EMG).
Usability and quality assessment of AMG and EMG monitoring | At the end of anesthesia (single assessment).
  Overall usability rating using a five-point Likert scale (1 = extremely poor, 5 = optimal) for AMG and EMG monitoring devices.
Incidence of postoperative respiratory complications | Through PACU discharge (approximately 1-2 hours after surgery).
  Number of participants experiencing respiratory complications (e.g., hypoxemia, airway obstruction, reintubation, or need for assisted ventilation) in the post-anesthesia care unit (PACU).
Perioperative changes in heart rate | From induction of anesthesia through PACU discharge.
  Heart rate (beats per minute, bpm) measured at predefined intraoperative and postoperative time points.
Perioperative changes in mean arterial pressure | From induction of anesthesia through PACU discharge
  Mean arterial pressure (mmHg) measured at predefined intraoperative and postoperative time points
Perioperative changes in oxygen saturation (SpO₂) | From induction of anesthesia through PACU discharge
  Oxygen saturation (SpO2), %) measured at predefined intraoperative and postoperative time points.
Perioperative changes in perfusion index | From induction of anesthesia through PACU discharge.
  Perfusion index (Unitless) measured at predefined intraoperative and postoperative time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedale - Università di Padova (Padua University Hospital), Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Aggregate, de-identified study results will be disseminated through peer-reviewed publications and conference presentations

REFERENCES:
- [Background] Carron M, Safaee Fakhr B, Ieppariello G, Foletto M. Perioperative care of the obese patient. Br J Surg. 2020 Jan;107(2):e39-e55. doi: 10.1002/bjs.11447. PMID 31903602
- [Background] Wedemeyer Z, Michaelsen KE, Jelacic S, Silliman W, Lopez A, Togashi K, Bowdle A. Accuracy and Precision of Three Acceleromyographs, Three Electromyographs, and a Mechanomyograph Measuring the Train-of-four Ratio in the Absence of Neuromuscular Blocking Drugs. Anesthesiology. 2024 Aug 1;141(2):262-271. doi: 10.1097/ALN.0000000000005051. PMID 38728090
- [Background] Naguib M, Brull SJ, Johnson KB. Conceptual and technical insights into the basis of neuromuscular monitoring. Anaesthesia. 2017 Jan;72 Suppl 1:16-37. doi: 10.1111/anae.13738. PMID 28044330
- [Background] Fuchs-Buder T, Romero CS, Lewald H, Lamperti M, Afshari A, Hristovska AM, Schmartz D, Hinkelbein J, Longrois D, Popp M, de Boer HD, Sorbello M, Jankovic R, Kranke P. Peri-operative management of neuromuscular blockade: A guideline from the European Society of Anaesthesiology and Intensive Care. Eur J Anaesthesiol. 2023 Feb 1;40(2):82-94. doi: 10.1097/EJA.0000000000001769. Epub 2022 Nov 15. PMID 36377554

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT07283354/Prot_SAP_000.pdf